CLINICAL TRIAL: NCT02381548
Title: A Phase 1 Study of AZD1775 in Combination With Belinostat in Relapsed and Refractory Myeloid Malignancies and Selected Untreated Patients With Acute Myeloid Leukemia
Brief Title: Phase I Trial of AZD1775 and Belinostat in Treating Patients With Relapsed or Refractory Myeloid Malignancies or Untreated Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Other - Adverse Events
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-00257; NCI-2015-00257 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MCC-12-07328; NCI-9853; 9853 (Other: University Health Network Princess Margaret Cancer Center LAO); 9853 (Other: CTEP); N01CM00100 (NIH); UM1CA186644 (NIH); UM1CA186716 (NIH)
Record Dates: First submitted 2015-03-05; First posted 2015-03-06 (Estimated); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia Post Cytotoxic Therapy; Blast Phase Chronic Myeloid Leukemia, BCR-ABL1 Positive; Myelodysplastic Syndrome; Recurrent Adult Acute Myeloid Leukemia; Recurrent Chronic Myeloid Leukemia, BCR-ABL1 Positive; Refractory Acute Myeloid Leukemia; Refractory Chronic Myeloid Leukemia, BCR-ABL1 Positive; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Blast Crisis; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — adavosertib; belinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (belinostat, WEE1 inhibitor AZD1775) (Experimental): Patients receive belinostat IV over 30-90 minutes QD on days 1-5 and 8-12 and WEE1 inhibitor AZD1775 PO QD on days 1-5 and 8-12. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Responding patients with CR, CRi, CRc, or CRm and do not go on to have stem cell transplant may only continue treatment for 3-4 additional courses after response.
  Interventions: Drug: Adavosertib; Drug: Belinostat; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Adavosertib — Given PO
  Other Names: AZD 1775; AZD-1775; AZD1775; MK 1775; MK-1775; MK1775
Drug: Belinostat — Given IV
  Other Names: Beleodaq; PXD 101; PXD-101; PXD101
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of WEE1 inhibitor AZD1775 and belinostat when given together in treating patients with myeloid malignancies that have returned after a period of improvement or have not responded to previous treatment or patients with untreated acute myeloid leukemia. WEE1 inhibitor AZD1775 and belinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) for a regimen combining WEE1 inhibitor AZD1775 (AZD1775) with belinostat in patients with refractory/relapsed acute myeloid leukemia (AML), chronic myeloid leukemia in blast crisis (CML-BC), or intermediate-2 or high-risk myelodysplastic syndrome (MDS), and selected previously untreated poor-prognosis patients with AML.

SECONDARY OBJECTIVES:

I. To describe the toxicities of this regimen. II. To observe and record anti-tumor activity. III. If responses are observed, to determine what relationship, if any, exists between such responses and tumor protein 53 (p53)/fms-related tyrosine kinase 3 (FLT3) mutational status.

IV. To describe pharmacokinetic (PK) interactions, if any, between AZD1775 and belinostat.

V. To test the feasibility of performing correlative studies involving leukemic blasts obtained pre-treatment and 24-hours post-treatment to determine if events associated with in vitro synergism (eg, down-regulation of phosphorylated [p]-Wee1 and p-checkpoint kinase 1 [Chk1]; dephosphorylation of cyclin-dependent kinase-like 1 [cdc2] at both tyrosine [Tyr]15 and threonine [Thr]14; increased expression of gamma H2A histone family, member X [H2A.X] and of p-histone H3 [HH3]) can be recapitulated following exposure to AZD1775 and belinostat in patients.

OUTLINE: This is a dose-escalation study.

Patients receive belinostat intravenously (IV) over 30-90 minutes once daily (QD) on days 1-5 and 8-12 and WEE1 inhibitor AZD1775 orally (PO) QD on days 1-5 and 8-12. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients achieving complete remission (CR), complete remission with incomplete blood count recovery (CRi), cytogenetic complete remission (CRc), or molecular complete remission (CRm) who do not go on to have stem cell transplant may only continue treatment for 3-4 additional courses after response.

After completion of study treatment, all patients are followed up for 30 days and responding patients are followed up every 2 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have one of the following, histologically or cytologically confirmed:

  * Acute myeloid leukemia (AML) [non- acute promyelocytic leukemia (APL) AML]

    * If previously treated:

      * AML that is relapsed or refractory to at least one prior line of therapy
    * If previously untreated, must meet all of the following:

      * >= 60 years of age
      * Secondary or therapy-related AML
      * Does NOT bear favorable cytogenetic and/or molecular features, eg, core-binding factor abnormalities, FLT3 Internal Tandem Duplication (FLT3-ITD) negative/NPM1 mutated, biallelic CCAAT/enhancer binding protein alpha (CEBPA) mutation without FLT3-ITD
  * Chronic myeloid leukemia blast crisis (CML-BC)

    * Relapsed or refractory to at least one Bcr-Abl-TKI-containing regimen
  * Myelodysplastic syndrome (MDS), must meet all of the following:

    * Higher risk MDS [intermediate-2 or high risk by the original International Prognostic Scoring System (IPSS)]
    * Relapsed, refractory, or intolerant to at least one prior line of therapy containing hypomethylating agents (deoxyribonucleic acid [DNA] methyltransferase inhibitors)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 50%)
* Total bilirubin =< 1.5 × upper limit of normal (ULN) for the laboratory unless resulting from hemolysis
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 × ULN for the laboratory
* Creatinine within normal limits for the laboratory OR creatinine clearance >= 60 mL/min/1.73 m^2 (estimated glomerular filtration rate [eGFR]) for patients with creatinine levels above the ULN for the laboratory
* Human immunodeficiency virus (HIV)-infected persons are eligible if they meet other eligibility criteria including the following:

  * No prior acquired immune deficiency syndrome (AIDS)-defining condition other than cluster of differentiation (CD)4+ cells nadir < 200/mm^3
  * Pre-leukemia CD4+ cell count >= 250/mm^3
  * Willing to adhere to antiretroviral therapy regimen with minimal overlapping toxicity and PK interactions with the experimental agents in this study; no zidovudine- and no ritonavir-containing regimens and no 3-drugs-in-1 pill regimens containing pharmacologic boosters are allowed; recommended regimens are integrase inhibitors combined with tenofovir and emtricitabine
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 4 months after completion of AZD1775 and belinostat administration
* Ability to swallow medication
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Clinical picture indicative of leukostasis or evidence of disseminated intravascular coagulopathy
* Other investigational agent within 3 weeks prior to initiation of study therapy
* Ongoing toxicities >= grade 2 from prior therapy
* Acute promyelocytic leukemia (APL, M3)
* Active central nervous system (CNS) leukemia
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD1775 or belinostat
* Stem cell transplant within previous 3 months prior to initiation of study therapy
* Major surgical procedures =< 28 days before beginning study treatment or minor surgical procedures =< 7 day before beginning study treatment; no waiting required after placement of a vascular access device
* Uncontrolled infection
* Pregnant or nursing; women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study therapy

  * Note: Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with AZD1775/belinostat
* Circulating blast count >= 50,000/uL within the week preceding enrollment
* Current candidacy for a potentially curative allogeneic stem cell transplant, unless declined
* Corrected QT (QTc) interval >= 450 ms (ie, grade 1 or higher) on electrocardiogram (ECG) prior to initiation of study treatment

  * If baseline QTc on screening ECG is >= 450 ms (ie, grade 1 or higher):

    * Check potassium and magnesium serum levels
    * Correct any identified hypokalemia and/or hypomagnesemia and repeat ECG to confirm QTc interval
  * For patients with baseline heart rate (HR) < 60 beats per minute (bpm) or > 100 bpm, manual measurement of QT interval by cardiologist is required, with Fridericia correction applied to that manual measurement to determine the QTc for eligibility consideration
  * Note: For patients with HR 60-100 bpm, manual measurement of QTc interval and use of Fridericia calculation is NOT required
* Any of the following related to risk of torsades de pointes and sudden cardiac death:

  * History of sustained ventricular tachycardia (VT), ventricular fibrillation (VF), torsades de pointes, or resuscitated cardiac arrest unless currently addressed with an implanted cardiac defibrillator
  * Concomitant treatment with an anti-arrhythmic agent to prevent or control arrhythmia; agents used for rate-control of atrial fibrillation are permitted provided that they are not prohibited due to potential drug interactions
  * Known congenital long QT syndrome
  * Second degree atrioventricular (AV) block type II, third degree AV block, or ventricular rate < 50 bpm or > 120 bpm
* Unstable angina, myocardial infarction or New York Heart Association (NYHA) class III/IV congestive heart failure within 30 days preceding study enrollment
* Ongoing or planned treatment with any of the following:

  * Atorvastatin
  * Strong inhibitors or inducers of cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4); as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product

    * If any of these agents have been used, patients must be off them for >= 2 weeks before starting study treatment
* Any known UGT1A polymorphism, heterozygous or homozygous
* History of prior therapy with belinostat or AZD1775
* Active gastrointestinal (GI) conditions that might predispose to drug intolerance or poor drug absorption
* Receiving any other therapies for cancer treatment (with the exception of gonadotropin-releasing hormone [GnRH] agonists for prostate cancer); Note: hydroxyurea is allowed before initiation of study treatment and for the first 5 days of study treatment
* Diagnosis or treatment for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, any in situ malignancy, or low-risk prostate cancer after curative therapy
* Medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk, interfere with the patient's participation in the study, or hinder evaluation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-08-18 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
Recommended phase 2 dose (RP2D) for the combination of WEE1 inhibitor AZD1775 and belinostat, defined as the dose in which =< 1 out of 6 patients at highest dose level below the maximally administered dose experience dose-limiting toxicities (DLTs) | 21 days
  Patients' treatment dosing level, dose modification, DLTs, and evaluability for DLTs will be listed and summarized by basic descriptive statistics (such as frequency and proportion). DLTs will be assessed according to the National Cancer (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0.

SECONDARY OUTCOMES:
Incidence of toxicity graded according to the National Cancer (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 30 days after completion of study treatment
  Adverse events (AEs) and serious AEs, dosing levels, treatment received, best clinical response, and demographics will be listed. Basic descriptive statistics will be used to summarize toxicities related to the study drugs by grade, and all toxicities, whether related or unrelated to the study drugs, and duration of response or stable disease to the combination therapy.
Response rate (complete remission [CR] + CR with incomplete blood count recovery [CRi] + cytogenetic CR [CRc] + molecular CR [CRm]) according to International Working Group and European Leukemia Net criteria | Up to 2 years
  The clinical best response rates will be calculated for each dose level, along with their corresponding 95% confidence intervals.
Duration of response (in patients with (complete remission [CR] + CR with incomplete blood count recovery [CRi] + cytogenetic CR [CRc] + molecular CR [CRm]) | From documentation of tumor response to disease progression or death, whichever occurs first, assessed up to 2 years
  Duration of response will be summarized by the first, second, and third quantiles and illustrated by a Kaplan-Meier plot.
Time to response | From registration to the time of documentation of tumor response, assessed up to 2 years
  Time to response will be summarized by the first, second, and third quantiles and illustrated by a Kaplan-Meier plot.
p53 and FLT3 mutation status | Up to 24 hours after first dose of study treatment
  A Chi-square test and a Fisher exact test will be used to determine if there is a significant association between clinical responses and p53/FLT3 mutational status. An ordinal regression (where best clinical responses are considered as an ordinal outcome variable) and a logistic regression (where best responses are dichotomized as yes or no responses) will be used to test the association between responses and p53/FLT3 mutational status, with adjustment of potential factors (e.g., dose level, age, sex).
Pharmacokinetic (PK) parameters (area under the curve [AUC], volume of distribution [Vd], peak concentration [Cmax], time to peak concentration [Tmax], and half-life [t1/2]) of belinostat | Day 1, course 1: pre-treatment, 5 minutes prior to the end of the belinostat infusion, 15 minutes (min), 30 min, 1 hour (hr), 2 hr, 4 hr, 6 hr, 8 hr, and 24 hr after the end of the belinostat infusion
  Will be calculated using standard non-compartmental methods and summarized as geometric mean and geometric coefficient of variation. Cmax and the times needed to reach these concentrations (tmax) will be assessed by inspection of the concentration versus time plots. The AUC will be calculated from time zero to infinity. Vd and t1/2 will also be calculated. To discover any potential PK interactions between the 2 agents, each PK parameter will be compared with each referenced PK parameter for those who receive single-agent at the same amount dose by a one-sample t-test.
PK parameters (area under the curve [AUC], volume of distribution [Vd], peak concentration [Cmax], time to peak concentration [Tmax], and half-life [t1/2]) of WEE1 inhibitor AZD1775 | Day 1, course 1: pre-treatment, and 30 min, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, and 24 hr after WEE1 inhibitor AZD1775 administration
  Will be calculated respectively using standard non-compartmental methods and summarized as geometric mean and geometric coefficient of variation. Cmax and the times needed to reach these concentrations (tmax) will be assessed by inspection of the concentration versus time plots. The AUC will be calculated from time zero to infinity. Vd and t1/2 will also be calculated. To discover any potential PK interactions between the 2 agents, each PK parameter will be compared with each referenced PK parameter for those who receive single-agent at the same amount dose by a one-sample t-test.
Changes in candidate biomarker levels (including p-Wee1, p-cdc2 and gamma-H2A.X) in bone marrow and/or blood samples | Baseline to 24 hours after first dose of study treatment
  Various paired t-tests will be used to determine if there is a significant change in each of the candidate biomarker between the pre- and 24-hour post-treatment assessments, in bone marrow samples and in blood samples. Various simple regression models will be used to check if there is an effect of potential factors (e.g., dose level, age, sex) on the change. The distribution of the change will be checked and if the data is highly skewed, then an appropriate data transformation will be conducted to satisfy the assumption of normality.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle A Shafer, Principal Investigator — University Health Network Princess Margaret Cancer Center LAO
Locations (2):
- United States (2):
  - Moffitt Cancer Center, Tampa, Florida
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia